CLINICAL TRIAL: NCT00986076
Title: Randomized Clinical Trial Evaluating Anti-inflammatory Effect of Low Molecular-Weight Heparin in Pediatric Cataract and Intraocular Lens Surgery
Brief Title: Clinical Trial on Anti-inflammatory Effect of Low-Molecular Weight Heparin in Pediatric Cataract Surgery
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Iladevi Cataract and IOL Research Center (Other)
Responsible Party: Viraj A. Vasavada, MS, Iladevi Cataract & IOL Research Centre
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 08-010
Record Dates: First submitted 2009-09-26; First posted 2009-09-29 (Estimated); Last update posted 2009-09-29 (Estimated); Status verified 2009-09

CONDITIONS: Inflammation
Keywords: Pediatric Cataract Surgery; Low-Molecular weight Heparin; Intraocular infusion; Anti-inflammatory effect
MeSH Terms: conditions — Inflammation | interventions — Enoxaparin; Hanks Balanced Salt Solution

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Enoxaparin infusion (Experimental): Congenital Cataract Surgery with IOL implantation
  Intraocular infusion of Enoxaparin
  Interventions: Drug: Enoxaparin
- Balanced Salt Solution Infusion (Placebo Comparator): Congenital Cataract Surgery with IOL implantation Intraocular infusion of Balanced Salt Solution
  Interventions: Drug: Balanced Salt Solution

INTERVENTIONS:
Drug: Enoxaparin — Enoxaparin 40 mg / 500 ml in Balanced Salt Solution
  Other Names: Clexane(Aventis)
  Arms: Enoxaparin infusion
Drug: Balanced Salt Solution — Intraocular infusion of Balanced Salt solution
  Other Names: BSS
  Arms: Balanced Salt Solution Infusion

SUMMARY:
The purpose of this study is to determine if intraocular infusion of low-molecular weight heparin (enoxaparin) influences postoperative inflammation following pediatric cataract surgery with intraocular lens (IOL) implantation.

DETAILED DESCRIPTION:
Despite advances in cataract surgery in children, postoperative inflammation is a significant complication following pediatric cataract surgery. Any drug that prevents or decreases this inflammation would be beneficial.

Heparin has anti-inflammatory and antiproliferative effects as well as anticoagulant properties. Several studies on animal and adult human eyes show that adding heparin to the irrigating solution during cataract surgery results in less disturbance of the blood-aqueous barrier and helps prevent posterior capsule opacification (PCO).

A prospective, randomized, controlled and masked study is mandatory to evaluate the anti-inflammatory effect of Low-molecular weight Heparin for pediatric cataract surgery

ELIGIBILITY:
Inclusion Criteria:

* Children (0-15 years) with congenital cataract scheduled for surgery with IOL implantation and informed consent from the parents/legal guardian

Exclusion Criteria:

* Preoperative: Associated ocular anomalies (uveitis, microphthalmos, persistent fetal vasculature, aniridia, glaucoma, iris coloboma), traumatic cataract
* Intraoperative: Inability to implant IOL in the capsular bag, intraoperative complications- iris trauma, vitreous disturbance, descemet's detachment

Max Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 23 (Actual)
Dates: Start 2008-03; Primary Completion 2009-04 (Actual); Study Completion 2009-09 (Actual)

PRIMARY OUTCOMES:
Anterior Segment Inflammation | 1 week

SECONDARY OUTCOMES:
Anterior Segment inflammation | 1 month, 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Viraj A Vasavada, MS, Principal Investigator — Iladevi Cataract & IOL Research Centre
Locations (1):
- Iladevi Cataract & IOL Research Centre, Ahmedabad, Gujarat, India

REFERENCES:
- [Background] Kruger A, Amon M, Abela-Formanek C, Schild G, Kolodjaschna J, Schauersberger J. Effect of heparin in the irrigation solution on postoperative inflammation and cellular reaction on the intraocular lens surface. J Cataract Refract Surg. 2002 Jan;28(1):87-92. doi: 10.1016/s0886-3350(01)00861-6. PMID 11777715
- [Background] Rumelt S, Stolovich C, Segal ZI, Rehany U. Intraoperative enoxaparin minimizes inflammatory reaction after pediatric cataract surgery. Am J Ophthalmol. 2006 Mar;141(3):433-7. doi: 10.1016/j.ajo.2005.08.020. PMID 16490487
- [Background] Wilson ME Jr, Trivedi RH. Low molecular-weight heparin in the intraocular irrigating solution in pediatric cataract and intraocular lens surgery. Am J Ophthalmol. 2006 Mar;141(3):537-8. doi: 10.1016/j.ajo.2005.11.012. No abstract available. PMID 16490502
- [Derived] Vasavada VA, Praveen MR, Shah SK, Trivedi RH, Vasavada AR. Anti-inflammatory effect of low-molecular-weight heparin in pediatric cataract surgery: a randomized clinical trial. Am J Ophthalmol. 2012 Aug;154(2):252-258.e4. doi: 10.1016/j.ajo.2012.02.021. Epub 2012 Apr 27. PMID 22541652